CLINICAL TRIAL: NCT04218292
Title: Dr. Amplatz Micro Plug - Post Market Clinical Follow-up (PMCF) Plan
Brief Title: Micro Plug Set - Post Market Clinical Follow-up (PMCF) Plan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KA Medical, LLC (Industry)
Collaborators: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF 24October2019; KAM-P4-21-01 (Other: Merit Medical Systems, Inc.)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Trauma Injury; Bleeding
MeSH Terms: conditions — Accidental Injuries; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Micro Plug Set — The Micro Plug Set is indicated for arterial embolization in the peripheral vasculature.

SUMMARY:
This is an observational, post market clinical follow-up (PMCF) intended to evaluate the residual risks of the Micro Plug Set which is intended for use during arterial embolization of the peripheral vasculature. This PMCF will collect data pertaining to any adverse events as well as the identification of any unanticipated risks up to the first 12 months following device implant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for arterial embolization in the peripheral vasculature.
* Subject is greater than 18 years of age

Exclusion Criteria:

* Subject is unable to give informed consent
* Subject is pregnant or breastfeeding
* Subject has allergy to nickel
* Patient requires neurologic or cardiac use of an occlusion device, contrary to the Micro Plug Set Instructions For Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring routine standard of care for peripheral embolization. Some of the patients will be liver cancer patients undergoing palliative treatment with SIRT who have a life expectancy that may be less than 12 months. Other patients may be treated for trauma or bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of serious device-related and procedure-related adverse events | 12 months
  Rate of serious device-related and procedure-related adverse events

SECONDARY OUTCOMES:
Rate of successful delivery of the device | 1 day
  Rate of successful delivery of the Micro Plug device to the intended position.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Pech, MD, Principal Investigator — University Hospital Magdeburg, Germany
Locations (1):
- University Hospital Magdeburg, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: No